CLINICAL TRIAL: NCT00220636
Title: Abilify (Aripiprazole) as an Adjunctive Treatment for Refractory Unipolar Depression
Brief Title: Abilify as an Adjunctive Treatment for Refractory Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLR-04-028
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2014-10

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depression; Depression; Unipolar Depression; Treatment Resistant Depression; Adjunctive treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): Aripiprazole 5 to 30 mg/day
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole dose ranging from 5 to 30 mg/day, augmenting antidepressant treatment. Aripiprazole is used as an augmenting medication on an open label basis for patients on antidepressant medication who continue to have depressive symptoms. This is an open label case series in which all subjects receive aripiprazole augmentation. There is no comparator group.
  Other Names: Abilify

SUMMARY:
This is a study of the effectiveness of adding Abilify (aripiprazole), an atypical antipsychotic medication, to ongoing selective serotonin reuptake inhibitor (SSRI) antidepressant treatment for depressed outpatients who are not responding fully to SSRI treatment alone. It is hypothesized that patients' functioning will improve after 12 weeks of treatment with Aripiprazole and SSRI medication.

DETAILED DESCRIPTION:
This is a pilot study of the effectiveness of adding Abilify (aripiprazole), an atypical antipsychotic medication, to ongoing selective serotonin reuptake inhibitor (SSRI) antidepressant treatment for depressed outpatients who are not responding fully to SSRI treatment alone. Fifteen subjects will be given aripiprazole in a flexible dosing schedule and followed for 12 weeks, while continuing their ongoing SSRI medication. Assessments of depressive symptoms, overall functioning, social functioning, and side effects will be completed. It is hypothesized that patients' functioning will improve after 12 weeks of treatment with Aripiprazole and SSRI medication.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of 18 and 70.
* Patients with a principal Diagnostic and Statistical Manual fourth edition (DSM-IV) diagnosis of Major Depressive Disorder, unipolar, nonpsychotic type
* Patients with a total of 14 or higher on the 17-item Hamilton Depression Scale at baseline
* Patients who have had treatment with an SSRI at an adequate dose (see Table for a minimum of 6 weeks (i.e. 6 wks at the dose defined as adequate in Table 2)
* Patients who agree to use acceptable method of birth control throughout the study

Exclusion Criteria:

* Patients with any of the following DSM-IV diagnoses: Delirium, Dementia, Amnestic, or other Cognitive Disorders. Bipolar Disorder or cyclothymia, Schizophrenia, Delusional (Paranoid) Disorders and Psychotic Disorders not elsewhere classified, Severe Borderline Personality Disorder, Anorexia Nervosa, or Bulimia.
* Patients who, within the past 6 months, met DSM-IV criteria for abuse of or dependence on any drug, including alcohol.
* Patients who are pregnant or nursing women.
* Patients who would pose a serious risk for suicide during the course of the study, as evidenced by one of the following: (a) report of having a specific plan for killing themselves, (b) a score of 3 or higher on the Hamilton Depression Rating Scale item #3 as rated by the treating clinician at Week 0, or (c) a suicide attempt within the last 6 months which required medical attention, such as an emergency room visit or which is considered by the treating physician to have been possibly life threatening
* Patients with unstable medical conditions such as untreated or uncontrolled hyperthyroidism, hypothyroidism, hypertension (defined as blood pressure>150/90), cardiovascular disease, diabetes, HIV (by report of patient).
* Patients with a history of seizures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hellerstein, MD, Principal Investigator — NY State Psychiatric Institute, and St. Luke's - Roosevelt Hospital Center
Locations (1):
- Depression Evaluation Service, NY State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Hellerstein DJ. Aripiprazole as an adjunctive treatment for refractory major depression. Prog Neuropsychopharmacol Biol Psychiatry. 2004 Dec;28(8):1347-8. doi: 10.1016/j.pnpbp.2004.06.016. No abstract available. PMID 15588762
- See also: Web Site for the Mood Disorders Research Program, with information about the study and the process of getting involved in research in general and specifically at our site — http://www.DepressionNY.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: aripiprazole augmentation treatment
Period: Overall Study
Arm/Group | Aripiprazole
Started | 15
Completed | 11
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS)
Description: Clinician rated measure of depression, mean score; this study used the 24 item version of the Hamilton Depression Rating Scale; item scores range from 0 to 4 on some items, 0 to 2 or 0 to 3 on other items; range of total score = 0 to 75, with higher score indicating worse depression Response (>50% decrease) Remission (score<=7) Outcome is the number of these subjects whose depression "responded" after treatment with aripiprazole, which means a 50% or greater decrease in Hamilton Depression Rating Scale scores at week 12.
Time Frame: 12 weeks
Population: Adults with treatment resistant depression, all subjects with data after baseline (14 of 15 subjects).
Measure: Number; unit: participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
participants | 7
Statistical Analysis 1: Comparison: Aripiprazole; Null hypothesis would be no change in the HDRS score pre- to post- treatment with aripiprazole; Test type: Superiority or Other; p < .001, t-test, 2 sided; df=13; t statistic = 4.7

2. Secondary Outcome: Clinical Global Impressions Improvement Scale (CGI)
Description: clinician rated improvement, score on CGI scale ranging from 1 (very much improved) to 7 (very much worse)
Time Frame: 12 weeks
Population: all subjects for whom data was available after beginning aripiprazole augmentation (14 of 15 subjects)
Measure: Mean (Standard Deviation); unit: units on CGI scale
Groups:
- Aripiprazole: aripiprazole augmentation treatment for treatment resistant depression
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
units on CGI scale | 2.8 (1.1)

3. Secondary Outcome: Change in Global Assessment of Functioning Scale (GAFS)
Description: Ranging from 0 to 100, with higher score indicating better global functioning. Outcome is the post-treatment GAFS score compared to the pre-treatment GAFS score.
Time Frame: baseline and 12 weeks
Population: All subjects (14/15) for whom data was available after starting aripiprazole augmentation
Measure: Mean (Standard Deviation); unit: points on GAFS scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
points on GAFS scale | 7.3 (4.7)
Statistical Analysis 1: Comparison: Aripiprazole; Null hypothesis would be no change in the GAFS score pre- to post- treatment with aripiprazole; Test type: Superiority or Other; p = .009, t-test, 2 sided; df=13; t statistic = -3.1

4. Secondary Outcome: Change in Beck Depression Inventory (BDI) Score
Description: 21 item patient rated assessment of depression symptoms, with item scores ranging from 0 to 3. Total BDI scores can range from 0 to 63, with higher scores indicating worse depression.
  Outcome is the subject's total BDI score post-treatment compared to the subject's total BDI score pre-treatment.
Time Frame: baseline and 12 weeks
Population: Number of participants for whom data was available after starting aripiprazole augmentation
Measure: Mean (Standard Deviation); unit: points on BDI scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 14
points on BDI scale | 4.2 (10.0)
Statistical Analysis 1: Comparison: Aripiprazole; Null hypothesis would be no change in the BDI score pre- to post- treatment with aripiprazole; Test type: Superiority or Other; p = .008, t-test, 2 sided; df=13; t statistic = 3.1

ADVERSE EVENTS:
Time Frame: 16 weeks, during and after the clinical trial
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=15)
fatigue (Nervous system disorders) | 8 (15)
nausea (Gastrointestinal disorders) | 7 (15)

LIMITATIONS AND CAVEATS:
Open label study without comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No